CLINICAL TRIAL: NCT03153774
Title: Assessments of Sarcopenia Prevalence in Chronic Heart Failure Patients and in Subjects Before Transcatheter Aortic Valve Implantation
Brief Title: Assessments of Sarcopenia Prevalence in Chronic Heart Failure Patients and in Subjects Before TAVI
Acronym: PRESAR-HF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHU-324; 2014-A00938-39 (Other: 2014-A00938-39)
Record Dates: First submitted 2017-05-05; First posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Sarcopenia; Chronic Heart Failure
Keywords: Sarcopenia; Heart failure (HF); The trans aortic valvular implantation (TAVI)
MeSH Terms: conditions — Sarcopenia; Heart Failure

STUDY DESIGN:
Masking Description: Open
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heart failure patients (Experimental): The main objective was to assess the prevalence of sarcopenia in chronic heart failure patients and in patients before the trans aortic valvular implantation.
  Interventions: Diagnostic Test: Assessment of sarcopenia prevalence
- TAVI patients (Experimental): The main objective was to assess the prevalence of sarcopenia in chronic heart failure patients and in patients before the trans aortic valvular implantation.
  Interventions: Diagnostic Test: Assessment of sarcopenia prevalence

INTERVENTIONS:
Diagnostic Test: Assessment of sarcopenia prevalence — Handgrip test, Bioimpedance analysis (Bodystat), 6-min walking test, Short physical performance battery (balance test, 4-min walking test, 5 times getting-up test), Biological markers test, Trans-thoracic echography, Electrocardiogram 12 leads, Palm gripping test

SUMMARY:
The main objective was to assess the prevalence of sarcopenia in chronic heart failure patients and in patients before the trans aortic valvular implantation.

The loss of muscle mass in chronic heart failure patients is a prognostic factor for sarcopenia. The purpose was to identify in these patients signs of sarcopenia for a better management.

DETAILED DESCRIPTION:
Age-related muscle loss, termed sarcopenia, affects 10% of elderly subjects aged 60-70 years and more than 30% above the age of 80. The concept of sarcopenia has been supported by the recent findings of muscular atrophy which was related to the decrease of protein synthesis because of the "anabolic resistance", affecting the muscular fibers type II. In fact, sarcopenia could be a consequence of chronic disease and not only an issue in the elderly people. The diagnosis is assessed by the weak muscle mass and the muscle strength and function. A description of these muscle parameters has been described in a study of 200 patients with NYHA class II-III and showed that 19,5 % have a decrease in muscle mass. They also showed that these patients have a lower functional ability. These findings prompted us to investigate the prevalence of sarcopenia in chronic heart failure subjects for a better management of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Major patients (>18 years)
* Men or women
* Hospitalized in pre- trans aortic valvular implantation assessment in the cardiology department of the university hospital centre of Clermont-Ferrand or
* Patients with chronic heart failure in charge in the hospital of Clermont-Ferrand or convalescence in the pneumocardiological clinic of Durtol

Exclusion Criteria:

* Patient not affiliated to social security
* Inability to understand the information consent letter
* Not having signed informed consent
* Has a mental or legal incapacitation and is unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-11-03 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Bioimpedance analysis data | at day 1
  Fat-free mass and body fat mass will be combined to report BMI in Kg/m2
Short physical performance battery | at day 1
  Balance test, 4-min walking test, 5 times getting-up test
Handgrip test | at day 1

SECONDARY OUTCOMES:
Blood draw for serum creatinine in umol/L | at day 1
  Measure of inflammation
CRP in mg/L | at day 1
  Measure of inflammation
platelets in Giga/L | at day 1
  Measure of inflammation
complete blood count CBC (white blood cells in Giga/L and red blood cells in Tera/L) | at day 1
  Measure of inflammation
urea in mmol/L | at day 1
  Measure of inflammation
albumin in g/L | at day 1
  Measure of inflammation
NT-ProBNP in ng/L | at day 1
  Measure of inflammation
Electrocardiogram | at day 1
  Parameter which may interfere with sarcopenia
Trans-thoracic echography | at day 1
  Parameter which may interfere with sarcopenia

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, Auvergne, France

REFERENCES:
- [Derived] Blanquet M, Massoulie G, Boirie Y, Guiguet-Auclair C, Mulliez A, Anker S, Boiteux MD, Jean F, Combaret N, Souteyrand G, Riocreux C, Pereira B, Motreff P, Rossignol P, Clerfond G, Eschalier R. Handgrip strength to screen early-onset sarcopenia in heart failure. Clin Nutr ESPEN. 2022 Aug;50:183-190. doi: 10.1016/j.clnesp.2022.05.019. Epub 2022 Jun 6. PMID 35871922
- [Derived] Eschalier R, Massoullie G, Boirie Y, Blanquet M, Mulliez A, Tartiere PL, Anker S, D'Agrosa Boiteux MC, Richard R, Jean F, Combaret N, Souteyrand G, Riocreux C, Pereira B, Motreff P, Stolt P, Rossignol P, Clerfond G. Sarcopenia in patients after an episode of acute decompensated heart failure: An underdiagnosed problem with serious impact. Clin Nutr. 2021 Jun;40(6):4490-4499. doi: 10.1016/j.clnu.2020.12.033. Epub 2021 Jan 9. PMID 33483182